CLINICAL TRIAL: NCT07356609
Title: Primary Care ERectile Function Outcome Registry for Men
Acronym: PERFORM
Status: Not yet recruiting | Type: Observational
Sponsor: Nabiqasim Industries (Pvt) Ltd (Industry)
Collaborators: Pakistan Society of Internal Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NQ/AP/SLR/Reg-007
Record Dates: First submitted 2026-01-08; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; male reproductive health; male sexual health
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PERFORM registry is a structured, real-world data platform designed to systematically capture patient characteristics, disease severity and treatment patterns of Erectile Dysfunction (ED) across Pakistan. By reflecting routine clinical practice, an ED registry provides valuable insights into the disease epidemiology, unmet needs, and variations in care across populations. It supports evidence-based decision-making, helps identifying early predictors, and inform guideline development, health policy, and personalized management strategies in male sexual health.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male above 18 years of age
2. Married
3. Diabetic
4. Patient reports erectile dysfunction (symptomatic).
5. Patient is eligible to be prescribed sildenafil by treating clinician.

Exclusion Criteria:

1. If at any other PDE-5 inhibitor (sildenafil, tadalafil, vardenafil, avanafil)
2. Concurrent use of organic nitrates (any form: glyceryl trinitrate, isosorbide mononitrate/dinitrate) - absolute contraindication
3. Recent or unstable cardiovascular disease

   * Myocardial infarction or stroke in last 3 months
   * Unstable angina
   * Uncontrolled arrhythmia or heart failure NYHA III-IV
   * Resting hypotension (SBP < 90 mmHg) or uncontrolled hypertension (SBP > 180 mmHg) per treating clinician
   * Known severe hepatic impairment or severe renal impairment on dialysis (if local clinician deems unsafe)
   * Known hypersensitivity to sildenafil or excipients
   * Concomitant use of potent CYP3A4 inhibitors (e.g., ritonavir) - unless clinician documents safe plan/dose adjustment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult Male ED patients
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Descriptive data of frequency, severity of ED in Pakistan | Baseline
  Prevalence
Descriptive data [age, income (derivative of socio-economic class), rural/urban population and occupation] | baseline
  Demographics

SECONDARY OUTCOMES:
Age of diabetes in ED patients | baseline
  Duration of diabetes in ED patients
Duration of ED | baseline
  Disease duration

IPD SHARING:
Plan to Share IPD: Undecided
Local sensitive data due to privacy concerns

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29650090/
- See also: Related Info — https://hospitals.aku.edu/pakistan/diseases-and-conditions/Pages/erectile-dysfunction.aspx
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29746858/
- See also: Related Info — https://uroweb.org/guidelines/sexual-and-reproductive-health/chapter/management-of-erectile-dysfunction
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40753504/
- See also: Related Info — https://www.scirp.org/reference/referencespapers?referenceid=2244060